CLINICAL TRIAL: NCT04368442
Title: Epidemiologic Evaluation and Clinical Outcomes for HER2-negative Metastatic Breast Cancer (MBC) Patients With Germline BRCA1 and 2 Pathogenic Mutation in Korea
Brief Title: Cohort Study of Patients With HER2-negative MBC and BRCA 1/2 Pathogenic Mutation
Acronym: BRCAm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, M.D., Ph.D., Division of hematology and oncology, Samsung Medical Center
Other Study IDs: 2019-06-027
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer Metastatic
Keywords: BRCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 1. DNA form the peripheral blood
  2. (optional) Extracted DNA from the FFPE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the prevalence germline pathogenic BRCA1/2 mutation in a large group of potential candidate of PARP inhibitors, among the unselected patients with HER2-negative unresectable locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, non-interventional study on the prevalence of germline pathogenic BRCA1/2 mutation (Blood) and somatic pathogenic BRCA1/2 mutation (Tissue, optional) in patients with HER2-negative unresectable locally advanced or metastatic breast cancer.

1. For the assessment of germline mutational status of BRCA1 and BRCA2, (1)Collect peripheral blood from each subject. (2) Extract DNA from the collected blood. (3)From the extracted DNA, germline BRCA1/2 mutational status will be assessed by next generation sequencing(NGS) using NGeneBioBRCAaccuTest®
2. For the assessment of somatic mutational status of BRCA1 and BRCA2, (1)Collect FFPE from about 100 subjects. (2) Extract DNA from the FFPE. (3)From the extracted DNA, somatic BRCA1/2 mutational status will be assessed by next generation sequencing(NGS) using NGeneBioBRCAaccuTest®
3. Collect variables on the patients and compare clinical outcomes (Overall survival, Invasive Disease-free survival, Distant Disease-free survival, Progression free survival) that can be affected by clinicopathologic characteristics and type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Histologically confirmed, unresectable locally advanced or metastatic breast invasive carcinoma
* Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer
* Germline mutational status of BRCA1 and/or BRCA2 can be known or unknown
* Signed written informed consent
* The patient is regarded as good candidate for active palliative management at time of enrollment. The patient with terminal cancer which is not appropriate for further endocrine treatment or chemotherapy cannot be enrolled to this study.

Exclusion Criteria:

* HER2 positive breast cancer
* Amenable to curative surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with HER2-negative unresectable locally advanced or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 583 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Length of time from the first date of each line of palliative endocrine treatment or chemotherapy until the date of the first documented progression of breast cancer or death of any cause,, assessed up to 60 months
  Progression free survival of each of palliative systemic treatment

SECONDARY OUTCOMES:
Overall survival 1 | Length of time from the date of first neoadjuvant chemotherapy or curative surgery until death for any cause,, assessed up to 60 months
  Overall survival from initial diagnosis
Overall survival 2 | Length of time from the first date of the first line of chemotherapy, assessed up to 60 months
  Overall survival from diagnosis of unresectable locally advanced/MBC
Disease-free survival | Length of time from the date of first neoadjuvant chemotherapy or curative surgery until the date of the first recurrence of breast cancer, diagnosis of second invasive cancer, or death for any cause whichever comes first, assessed up to 60 months
  Invasive Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: YEON HEE PARK, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea